CLINICAL TRIAL: NCT02693015
Title: Impact of Time to Coronary Angiography on Survival for NSTEMI: an Observation Study Using a Nationwide Registry
Brief Title: Impact of Time to Coronary Angiography on Survival for NSTEMI
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Dr Christopher Gale, Associate Professor, University of Leeds
Other Study IDs: Time to coronary angiography
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Non ST-elevation Myocardial Infarction
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to investigate the extent to which the time to angiography impacts on survival in patients hospitalised with NSTEMI.

DETAILED DESCRIPTION:
The use of an invasive strategy for the management of NSTEMI according to estimated risk of 6 month mortality is recommended by international guidelines. NSTEMI appropriate for coronary angiography (and percutaneous intervention) have better outcomes compare with NSTEMI who are medically managed. Whilst the national and international guidelines recommend that the timing of (in-hospital) coronary angiography (<24, 24-72, 72-96 and <96 hours) is based upon estimated clinical risk (using the GRACE risk score) there is scientific and clinical uncertainty as to the incremental benefit that more urgent invasive treatments strategies have over and above that of delayed strategies. Moreover, the investigators recent research has shown that in the UK, may NSTEMI (eligible) for coronary angiography fail to achieve care according to the recommended time thresholds, and this is associated with potentially avoidable premature death.

This study aims to investigate the extent to which the time to angiography impacts on survival in patients hospitalised with NSTEMI. It will characterise patients according to their estimated risk of death, their time to angiography, and associated outcomes. The investigators anticipate that this observational study will provide Level B evidence for the benefits of the timing of an invasive strategy according to the GRACE risk score. The investigators are aware that the NICE guidelines for the management of acute chest pain are to be updated in 2016.

ELIGIBILITY:
Inclusion Criteria:

* The target population will be all patients aged 18 to 100 years recorded within MINAP from 2004 to 2013 who have been hospitalised with NSTEMI and received coronary angiography.

Exclusion Criteria:

* Age below 18 or above 100 or age missing
* Diagnosis not NSTEMI
* Patients who did not receive coronary angiography - as this is the investigators explanatory variable

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises 725,860 patients hospitalised for acute myocardial infarction and entered into the Myocardial Ischaemia National Audit Project (MINAP) database between April 2004 and March 2013.
Sampling Method: Non-Probability Sample
Enrollment: 235986 (Actual)
Dates: Start 2004-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 30-day mortality since hospitalisation
Mortality | 1-year mortality since hospitalisation